CLINICAL TRIAL: NCT07030400
Title: Predictors of Health-Related Quality of Life in Adults With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: Predictors of Health-Related QOL in Adults With CLL or Small Lymphocytic Lymphoma
Status: Recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network); AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: MCC-23558
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Small Lymphocytic Lymphoma (SLL); Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bruton's tyrosine kinase inhibitor treatment: Patients treated with a Bruton's tyrosine kinase inhibitor.
  Interventions: Drug: Bruton's tyrosine kinase inhibitor
- B-Cell Lymphoma 2 Protein Inhibitor treatment: Patients treated with a B-Cell Lymphoma 2 Protein Inhibitor.
  Interventions: Drug: B-Cell Lymphoma 2 Protein Inhibitor

INTERVENTIONS:
Drug: Bruton's tyrosine kinase inhibitor — BTKi
  Groups: Bruton's tyrosine kinase inhibitor treatment
Drug: B-Cell Lymphoma 2 Protein Inhibitor — BCL2i
  Groups: B-Cell Lymphoma 2 Protein Inhibitor treatment

SUMMARY:
The study aims to improve our understanding of how quality of life, fatigue, and symptoms change over 2 years when participants are treated for chronic lymphocytic leukemia or small lymphocytic lymphoma. We will compare two types of treatment to help future patients with chronic lymphocytic leukemia or small lymphocytic lymphoma know what to anticipate.

ELIGIBILITY:
Inclusion Criteria:

* All patients with pathology-confirmed diagnoses of CLL who are within seven days of starting treatment with a BTKi +/- an anti-CD 20 monoclonal antibody or BCL2i with Obinutuzumab treatment will be included.
* Subjects must be able to read and speak English or Spanish at the 8th grade level.

Exclusion Criteria:

* Patients with dementia, traumatic brain injury, or individuals with central nervous system involvement of their leukemia will be excluded from study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18 years of age and older with a diagnosis of CLL/SLL who are starting treatment with either a Bruton tyrosine kinase inhibitor +/-an anti-CD 20 monoclonal antibody or a B cell lymphoma 2 inhibitor (BCL2i) with Obinutuzumab.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Health Related Quality of Life (HRQOL) | Up to 2 years
  Compare the differences in HRQOL scores measured by the Functional Assessment of Cancer Therapy Leukemia version for patients receiving BTKi, and BCL2i within 7 days of beginning treatment and at days 30,60, 90, 180, 1 year, 1.5 years, and 2 years following initiation of treatment.
HRQOL predictors | Up to 2 years
  Investigators will test how age, comorbidity, fatigue, symptoms, and disease characteristics are related to the slope of HRQOL in separate models.
Interactions with treatment | Up to 2 years
  Three models will assess interactions between treatment and age, comorbidity, and fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tinsley-Vance, PhD, APRN, AOCN, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided